CLINICAL TRIAL: NCT05474508
Title: Effects of Diaphragmatic Breathing With and Without Aerobic Exercise on Stress, Fatigue and Sleep Quality Among Post Postpartum Women
Brief Title: Effects of Diaphragmatic Breathing With and Without Aerobic Exercise on Stress, Fatigue and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0531
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Stress; Fatigue; Sleep
Keywords: Diaphragmatic Breathing; Exercise; Fatigue; Postpartum; Stress
MeSH Terms: conditions — Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic breathing along with aerobic exercises (Experimental): Experimental Group (Group A) will receive both aerobic exercises and diaphragmatic breathing exercise. Exercise programs will consist of 1 set of contractions per day and each set will include 30 repetitions for 6 weeks. Exercise protocol consist of at least 150 minutes of moderate-intensity aerobic activity every week dividing the 150 minutes into 30-minute workouts on 5 days of the week or into smaller 10-minute sessions throughout each day will be carried out for 6 weeks
  Interventions: Other: Diaphragmatic breathing; Other: Aerobic exercises
- Diaphragmatic breathing only without aerobic exercises (Active Comparator): Active comparator (Group B) will receive only diaphragmatic breathing exercises. Exercise programs will consist of 1 set of contractions per day and each set will include 30 repetitions for 6 weeks.
  Interventions: Other: Diaphragmatic breathing

INTERVENTIONS:
Other: Diaphragmatic breathing — Exercise programs will consist of 1 set of contractions per day and each set will include 30 repetitions for 6 weeks.
Other: Aerobic exercises — Exercise protocol consist of at least 150 minutes of moderate-intensity aerobic activity every week dividing the 150 minutes into 30-minute workouts on 5 days of the week or into smaller 10-minute sessions throughout each day will be carried out for 6 weeks.
  Arms: Diaphragmatic breathing along with aerobic exercises

SUMMARY:
The puerperium is a critical phase for women , not only does it have a significant impact on the mental and physical health of fresh mothers, but it can also be one of the most stressful moments in a woman's life .Serious psycho- social problems, including fatigue, depression, and stress, have been reported that occurred during the postpartum period. Diaphragm breathing method (DBE).DBE, also known as Diaphragmatic Breathing or Deep Breathing, is an effective holistic mind body workout for coping with stress and physical and mental conditions.Postpartum fatigue is considered the foremost common issue that postnatal ladies stand up to when they move to motherhood.postpartum fatigue is described as sentiments of fatigue,suffocation and diminishes in physical and mental capacity.

This study will be a randomized clinical trial. Sample will be collected through convenient sampling technique.Randomization will be done through lottery method and patients will be divided into two groups. Group A will receive both aerobic exercises and diaphragmatic breathing exercise. B will receive only diaphragmatic breathing exercise. Data will be collected before and after treatment .data will be analyzed through SPPS 25.

DETAILED DESCRIPTION:
The puerperium is a critical phase for women , not only does it have a significant impact on the mental and physical health of fresh mothers, but it can also be one of the most stressful moments in a woman's life .Serious psycho- social problems, including fatigue, depression, and stress, have been reported that occurred during the postpartum period. As a result, postpartum psychological problems can affect the new mother's ability to care for children and affect her quality of life. Sleep problems, such as poor sleep quality and sleep disturbance, often occur in perinatal and postnatal women.Studies have shown that non- pharmacological interventions for postoperative pain reduce pain intensity. One of these non-pharmacological methods is the diaphragm breathing method (DBE).DBE, also known as Diaphragmatic Breathing or Deep Breathing, is an effective holistic mind body workout for coping with stress and physical and mental conditions.Postpartum fatigue is considered the foremost common issue that postnatal ladies stand up to when they move to motherhood.postpartum fatigue is described as sentiments of fatigue,suffocation and diminishes in physical and mental capacity.

This study will be a randomized clinical trial. Sample will be collected through convenient sampling technique.Randomization will be done through lottery method and patients will be divided into two groups. Group A will receive both aerobic exercises and diaphragmatic breathing exercise. Exercise programs will consist of 1 set of contractions per day and each set will include 30 repetitions for 6 weeks. Exercise protocol consist of at least 150 minutes of moderate-intensity aerobic activity every week dividing the 150 minutes into 30-minute workouts on 5 days of the week or into smaller 10-minute sessions throughout each day will be carried out for 6 weeks.Group B will receive only diaphragmatic breathing exercise. Exercise programs will consist of 1 set of contractions per day and each set will include 30 repetitions for 6 weeks. Data will be collected before and after treatment .data will be analyzed through SPPS 25.

ELIGIBILITY:
Inclusion Criteria:

* Women with age group of 20- 40 were included in study.
* Women who had Vaginal or c section delivery were included in study.
* Women with no postnatal complications were included in study.

Exclusion Criteria:

* Women who had a major operation within the last 3years were excluded.
* Women who had chronic issues i.e diabetes, hypertension were excluded.
* Women who had a history of psychiatric disorders were excluded.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 48 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Perceived stress scale | 6 Weeks
  The Perceived Stress Scale is the most often used psychometric tool for assessing stress sensitivity. It is an assessment of how difficult things in one's life are perceived to be.
Pittsburgh sleep quality index | 6 Weeks
  The PSQI is a 19-item, self-reported questionnaire used to assess sleep quality.
Fatigue severity scale | 6 Weeks
  The FSS assessment has nine statements that assess the intensity of your tiredness symptoms. Read the information and mark a value from 1 to 7 depending on the how precisely it depicts your situation over the last week and how much you disagree or agree that now the claim pertains to yourself

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, gynae ward, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buckley SJ. Executive Summary of Hormonal Physiology of Childbearing: Evidence and Implications for Women, Babies, and Maternity Care. J Perinat Educ. 2015;24(3):145-53. doi: 10.1891/1058-1243.24.3.145. PMID 26834435
- [Background] Asadi M, Noroozi M, Alavi M. Factors Affecting Women's Adjustment to Postpartum Changes: A Narrative Review. Iran J Nurs Midwifery Res. 2020 Nov 7;25(6):463-470. doi: 10.4103/ijnmr.IJNMR_54_20. eCollection 2020 Nov-Dec. PMID 33747834
- [Background] Kolovetsiou-Kreiner V, Moertl MG, Papousek I, Schmid-Zalaudek K, Lang U, Schlembach D, Cervar-Zivkovic M, Lackner HK. Maternal cardiovascular and endothelial function from first trimester to postpartum. PLoS One. 2018 May 21;13(5):e0197748. doi: 10.1371/journal.pone.0197748. eCollection 2018. PMID 29782509
- [Background] Umazume T, Yamada T, Yamada S, Ishikawa S, Furuta I, Iwano H, Murai D, Hayashi T, Okada K, Morikawa M, Yamada T, Ono K, Tsutsui H, Minakami H. Morphofunctional cardiac changes in pregnant women: associations with biomarkers. Open Heart. 2018 Jul 16;5(2):e000850. doi: 10.1136/openhrt-2018-000850. eCollection 2018. PMID 30057771
- [Background] Bett GC. Hormones and sex differences: changes in cardiac electrophysiology with pregnancy. Clin Sci (Lond). 2016 May 1;130(10):747-59. doi: 10.1042/CS20150710. PMID 27128800